CLINICAL TRIAL: NCT06325735
Title: Combined Systemic Inflammatory Indices and Their Impact on Birth Weight: A Prospective Observational Study.
Brief Title: Combined Systemic Inflammatory Indices and Birth Weight
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Marco La Verde, Researcher, University of Campania Luigi Vanvitelli
Other Study IDs: 98
Record Dates: First submitted 2024-03-10; First posted 2024-03-22 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Systemic Inflammation Markers; Birth Weight; Combined Systemic Inflammatory Indices
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- full term pregnancy: Total Participants: The study included full-term pregnant women.
  Exclusion Criteria: Participants were carefully selected, excluding those with specific conditions that could confound the study results. These conditions included gestational and pregestational diabetes, chronic hypertension, gestational hypertension, pre-eclampsia/eclampsia, intrauterine fetal growth restriction, preterm delivery, multiple pregnancies, and prenatally detected fetal abnormalities.
  Interventions: Diagnostic Test: None intervention

INTERVENTIONS:
Diagnostic Test: None intervention — None intervention, observational study

SUMMARY:
The study aimed to explore the complex relationship between various systemic inflammatory indices and birth weight

DETAILED DESCRIPTION:
The research was structured as a prospective observational study. It was conducted at a second-level University Hospital over the period from December 2019 to February 2021.

Participants:

Blood samples were collected at hospital admission. These samples were used for a complete blood count, focusing specifically on deriving systemic inflammatory indices.

The primary inflammatory indices studied were Neutrophil-to-Lymphocyte Ratio (NLR), Platelet-to-Lymphocyte Ratio (PLR), and Monocyte-to-Lymphocyte Ratio (MLR).

The birth weight was registered.

ELIGIBILITY:
Inclusion Criteria:

* physiological Full-term pregnancies

Exclusion Criteria:

* gestational diabetes
* pregestational diabetes
* Chronic Hypertension
* Gestational Hypertension
* Preeclampsia
* Eclampsia
* Intrauterine Fetal Growth Restriction
* Preterm Delivery
* Multiple Pregnancies
* Fetal malformations

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population comprised full-term pregnant women. These participants were likely to represent a diverse range of ages and backgrounds, typical of a general pregnant population at a second-level University Hospital.
  Health Status: The women included were in generally good health, with full-term, uncomplicated pregnancies. This was ensured by the rigorous exclusion of any pregnancies affected by significant health issues such as diabetes, hypertension, and other specified conditions.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Systemic inflammatory indices and birth weight | 3 months
  investigate the correlation between systemic inflammatory indices and birth weight in full-term pregnancies

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli studi della Campania "Luigi Vanvitelli"- OB & Gyn -, Napoli, Italia, Italy

IPD SHARING:
Plan to Share IPD: No